CLINICAL TRIAL: NCT06611085
Title: The Effect of Cold Application, Vibration and Vibrating Ice on Pain, Fear and Satisfaction Level in Children Aged 7-12 Years Who Underwent Blood Glucose Level Measurement
Brief Title: Cold Application, Vibration and Vibrating Ice on Pain, Fear and Satisfaction Level in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Atiye Karakul, Assoc. Prof., Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-8-17
Record Dates: First submitted 2024-09-23; First posted 2024-09-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Fear; Pain; Satisfaction
Keywords: fear; pain; satisfaction
MeSH Terms: conditions — Pain; Personal Satisfaction | interventions — Vibration

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cold application group (Experimental): The index finger of the child will be used in the cold application group. In this group, cold application will be performed by placing the index finger of the designated hand on a 10 x 10 cm ice pack for 30 seconds and then removing the ice pack immediately.
  Interventions: Other: cold application group
- vibration group (Experimental): The middle finger of the child will be used in the vibration group. In this group, vibration was applied by targeting the tip of the middle finger area using a vibrator device measuring 2x1x3 cm. The insertion of the needle will coincide with the application of the vibration stimulation.
  Interventions: Other: vibration group
- vibration and ice group (Experimental): In the vibration and ice group, cold and vibration stimulation will be applied to the child simultaneously. The ring finger of the designated hand was placed on a 10x10 cm ice pack for 30 seconds and subjected to cold application. Simultaneously, vibration stimulation will be applied to the tip of the middle finger area using a vibrator device with dimensions of 3x1 cm and 2x1 cm. After 30 seconds, the ice bag will be removed and the lancet pen will be adjusted for drilling from the fingertip while vibration stimulation continues.
  Interventions: Other: vibration and ice group
- Control (No Intervention): After determining the hands for intervention and control, measurement will be made according to the clinical routine for the first control. In clinical routine practice, in the measurement of blood glucose level, a puncture is performed with a lancet pen, then the first blood is wiped off and the second blood is measured with a glucometer.

INTERVENTIONS:
Other: cold application group — The index finger of the child will be used in the cold application group. In this group, cold application will be performed by placing the index finger of the designated hand on a 10 x 10 cm ice pack for 30 seconds and then removing the ice pack immediately.
  Arms: cold application group
Other: vibration group — The middle finger of the child will be used in the vibration group. In this group, vibration was applied by targeting the tip of the middle finger area using a vibrator device measuring 2x1x3 cm. The insertion of the needle will coincide with the application of the vibration stimulation.
  Arms: vibration group
Other: vibration and ice group — In the vibration and ice group, cold and vibration stimulation will be applied to the child simultaneously. The ring finger of the designated hand was placed on a 10x10 cm ice pack for 30 seconds and subjected to cold application. Simultaneously, vibration stimulation will be applied to the tip of the middle finger area using a vibrator device with dimensions of 3x1 cm and 2x1 cm. After 30 seconds, the ice bag will be removed and the lancet pen will be adjusted for drilling from the fingertip while vibration stimulation continues.
  Arms: vibration and ice group

SUMMARY:
The aim of this study was to determine the effects of cold application, vibration and vibrating ice on pain, fear and satisfaction levels in children aged 7-12 years who underwent blood glucose level measurement.The population of the study will consist of children aged 7-12 years who receive treatment and care in the pediatric ward of the Ministry of Health, University of Health Sciences, Izmir Tepecik Training and Research Hospital between July 2024 and July 2025. Descriptive Information Form, Child Fear Scale, Numerical Pain Scale and Child Satisfaction Scale will be used to collect the research data.

DETAILED DESCRIPTION:
Pain and painful experiences make the child more vulnerable to pain. Since it is not possible to eliminate the feeling of pain in pediatric patients, effective pain management has an important place . This study aimed to determine the effects of cold application, vibration and vibrating ice on pain, fear and satisfaction levels in children aged 7-12 years who underwent blood glucose level measurement.The population of the study will consist of children aged 7-12 years who receive treatment and care in the pediatric ward of the Ministry of Health, University of Health Sciences, Izmir Tepecik Training and Research Hospital between July 2024 and July 2025. Collection of Research Data The study will be started after ethics committee approval and written institutional authorisation.

Data will be collected before blood glucose measurement according to the clinical routine and the time of blood glucose measurement of the child. In the collection of data, pediatric patients admitted to the paediatric ward and their parents who meet the inclusion criteria of the study and agree to participate in the study will be informed about the purpose of the study and the study and their verbal and written permissions will be obtained.

* Data collection forms (Descriptive Information Form, Fear Scale) will be applied to the children and parents in the sample group. Fear assessment of the child will be done by the child, nurse and parent.
* The hand to be used for intervention will be determined by lottery. Cards labelled right and left will be prepared and the child will be asked to draw from the envelope in a closed manner.
* After determining the hands for intervention and control, measurements will be made according to the clinical routine for the first control. In clinical routine practice, in the measurement of blood glucose level, a puncture is performed with a lancet pen, then the first blood is wiped off and the second blood is measured with a glucometer.
* Intervention:
* The index finger of the child will be used in the cold application group. In this group, cold application will be performed by placing the index finger of the designated hand on a 10 x 10 cm ice pack for 30 seconds and then removing the ice pack immediately.
* In the vibration group, the middle finger of the child will be used. In this group, vibration was applied by targeting the tip of the middle finger area using a vibrator device measuring 2x1x3 cm. The insertion of the needle will coincide with the application of the vibration stimulation.
* In the vibration and ice group, cold and vibration stimulation will be applied to the child simultaneously. The ring finger of the designated hand was placed on a 10x10 cm ice pack for 30 seconds and subjected to cold application. Simultaneously, vibration stimulation will be applied to the tip of the middle finger area using a vibrator device with dimensions of 3x1 cm and 2x1 cm. After 30 seconds, the ice bag will be removed and the lancet pen will be adjusted for drilling from the fingertip while vibration stimulation continues.

After blood glucose measurement, Fear Scale, Numerical Pain Scale and Child Satisfaction Scale will be applied after each non-pharmacological intervention. Fear and pain assessment of children will be done by the child, nurse and parent.

ELIGIBILITY:
Inclusion Criteria:

* To be between 7-12 years old
* Blood glucose monitoring of the child
* Measurement of blood glucose at least 4 times a day
* Volunteering to participate in the study

Exclusion Criteria:

* Having another chronic disease
* Use of painkillers
* Communication, mental or neurological problems
* Having a skin condition on the finger

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
fear level | 1 day
  Fear Scale: It was developed by Thurillet et al. to evaluate children's fears based on self-report of children aged 4-12 years. Turkish validity and reliability study was conducted by Tavşan et al. The scale consists of six facial expressions. The scale grades fear with a score ranging from 0 to 10 (gradually graded two by two) consistent with pain rating scales. The first facial expression indicates that there is no fear, the fear increases from right to left, and the sixth facial expression indicates that the level of fear is the highest.
pain level | 1 day
  Numerical Pain Scale, this method, which aims to determine the severity of pain, aims to explain the patient's pain with numbers. In numerical scales, absence of pain (0) is evaluated as unbearable pain.
Satisfaction level | 1 day
  The Child Satisfaction Scale was developed by the researchers in line with the literature in a way that pediatric patients can easily understand. The numbers between 0 and 10 were placed on a horizontal line by circling the point corresponding to the satisfaction of the children with the education given. In the scale, 0 points means 'not satisfied at all' and 10 points means 'extremely satisfied'.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Tarsus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Hayek, A. A., Robert, A. A., Babli, S., Almonea, K. ve Al Dawish, M. A. (2017). Fear of Self-Injectingand Self-TestingandtheRelated Risk Factors in AdolescentswithType 1 Diabetes: A Cross-SectionalStudy. DiabetesTherapy, 8(1). doi:10.1007/s13300-016-0221-8
- [Background] Andersson V, Bergman S, Henoch I, Simonsson H, Ahlberg K. Pain and pain management in children and adolescents receiving hospital care: a cross-sectional study from Sweden. BMC Pediatr. 2022 May 5;22(1):252. doi: 10.1186/s12887-022-03319-w. PMID 35513880
- [Background] Bergomi P, Scudeller L, Pintaldi S, Dal Molin A. Efficacy of Non-pharmacological Methods of Pain Management in Children Undergoing Venipuncture in a Pediatric Outpatient Clinic: A Randomized Controlled Trial of Audiovisual Distraction and External Cold and Vibration. J Pediatr Nurs. 2018 Sep-Oct;42:e66-e72. doi: 10.1016/j.pedn.2018.04.011. Epub 2018 May 1. PMID 29728296
- [Background] Hanberger L, Tallqvist E, Richert A, Olinder AL, Forsner M, Morelius E, Nilsson S. Needle-Related Pain, Affective Reactions, Fear, and Emotional Coping in Children and Adolescents With Type 1 Diabetes: A Cross-Sectional Study. Pain Manag Nurs. 2021 Aug;22(4):516-521. doi: 10.1016/j.pmn.2021.01.007. Epub 2021 Feb 25. PMID 33640255
- [Background] Yu Z, Zhou Y, Xu X, Lin L, Le Q, Gu Y. Pharmacological and non-pharmacological interventions in management of peripheral venipuncture-related pain: a randomized clinical trial. BMC Pediatr. 2023 Feb 3;23(1):58. doi: 10.1186/s12887-023-03855-z. PMID 36737707
- [Background] Yaz SB, Basdemir S, Gectan E. The effect of vibrating cold application and puppet use on pain and fear during phlebotomy in children: A randomized controlled study. J Pediatr Nurs. 2024 Jan-Feb;74:77-84. doi: 10.1016/j.pedn.2023.11.018. Epub 2023 Nov 28. PMID 38029689